CLINICAL TRIAL: NCT01243476
Title: Multicenter, Randomized, Double-blind, Phase III Study of REVLIMID (Lenalidomide) Versus Placebo in Patients With Low Risk Myelodysplastic Syndrome (Low and Intermediate-1 IPSS) With Alteration in 5q- and Anemia Without the Need of Transfusion.
Brief Title: Study of REVLIMID (Lenalidomide) Versus Placebo in Patients With Low Risk Myelodysplastic Syndrome
Acronym: SINTRA-REV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fundación General de la Universidad de Salamanca (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SINTRA-REV; 2009-013619-36 (EudraCT Number)
Record Dates: First submitted 2010-11-17; First posted 2010-11-18 (Estimated); Last update posted 2023-02-15 (Actual); Status verified 2023-01

CONDITIONS: Myelodysplastic Syndrome
Keywords: myelodysplastic syndrome; 5q deletion; anemia; lenalidomide; red blood cells transfusion
MeSH Terms: conditions — Myelodysplastic Syndromes; Anemia | interventions — Lenalidomide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- lenalidomide (Experimental): Experimental treatment branch with Lenalidomide 5 mg/day (oral use)
  Interventions: Drug: Lenalidomide
- placebo (Placebo Comparator): Placebo branch (oral use)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Lenalidomide — Treatment with Revlimid (lenalidomide), oral use, 5 mg daily during study treatment (104 weeks).
  Other Names: Revlimid 5 mg
  Arms: lenalidomide
Other: Placebo — Placebo, oral use, daily during study treatment (104 weeks)
  Arms: placebo

SUMMARY:
Trial Design:

This clinical trial is a phase III multicenter, randomized, double blind and controlled with placebo trial and with two arms designed to assess the efficiency and toxicity of the scheme Lenalidomide versus observation in a series of 60 patients with low risk myelodysplastic syndrome associated to 5q deletion with anemia (Hb≤12g/dL) but without the need of transfusion. Patients are randomized in the study in a 2:1 ratio. They will receive treatment for 104 weeks until progression of the disease, which implies that the patient suffering from anemia due to myelodysplastic syndrome requires transfusion of at least 2 UCH/56 days (2 months) with a minimum follow up of 112 days (4 months), or unacceptable toxicity.

Disease:

Low risk myelodysplastic syndrome associated to the loss of 5q without transfusion requirements.

Total number of patients:

In total 60 patients will be included, 40 assigned to the treatment branch and 20 to the placebo branch.

Calendar:

First patient first visit: February 2010, and Last patient last visit expected in February 2016. (Recruitment was initially expected to take place over a period of 24 months and was expected to be finished in February 2012, but due to low rate of recruitment it was extended until the population sample is included in the trial).

DETAILED DESCRIPTION:
General summary of myelodysplastic syndrome with alteration in 5q. Myelodysplastic syndromes (MDS) are a very heterogenic group of diseases characterized by the presence of morphologic features of dyshemopoiesis in bone marrow (BM) and in peripheral blood (PB), which is translated into an inefficient hematopoiesis. This will lead to the concomitant development of peripheral cytopenias which will be the cause of complications in these patients and, in most cases, the cause of death. In addition, these patients have an increased risk of developing acute leukemia, and this risk increases with the progression of the disease.MDS represents an incurable disease with standard treatments with a quite variable survival mean ranging from 3 months to 15 years depending on the number of blasts, the number of cytopenias and the type of cytogenetic disorders2. The sole curative treatment of the MDS is the allogenic transplant of hematopoietic progenitors but this option is only available for a 5% of the patients with MDS.

Lenalidomide, initially known as CC-5013, is an analogue of the immunomodulator Drug Thalidomide (Thalidomid®; Pharmion Corp., Boulder, CO, USA), which was the first drug with anti-angiogenic and immunomodulator properties investigated in MDS. Lenalidomide has, as well as thalidomide, a broad array of potential activities against dysplastic cells, not fully known, among which we find immunomodulator and non-immunomodulator properties (anti-angiogenic effect, anti-proliferative and pro-apoptotic). The greater advantage of Lenalidomide in comparison with thalidomide is that the former is between 50 and 2000 times stronger tan thalidomide in what respects to its immunomodulator effects. And moreover, the toxic profile of Lenalidomide seems lower than that of its analogue; Thalidomide.

There is no treatment indication on the present times for patients with low risk MDS associated to the loss of 5q without transfusion dependent anemia. The results with Lenalidomide are highly promising for patients with low risk MDS associated to the loss of 5q when (it has so been tested) there is red blood cells transfusion dependent anemia. In this sense, the proposal consists on being able to state that treatment with Lenalidomide can be efficient from diagnose preventing CH transfusions with an acceptable toxicity.

In this sense, the present study has the intention to treat early patients with low-risk MDS associated to the loss of 5q with a view to prevent CH transfusion. Therefore, we could extend in these patients the time until CH transfusion and even assess the possibility of eradicating the disease at a cytogenetic/morphologic level. In the present trial and given the characteristics of the patients, we have chosen the option of supplying Lenalidomide at a dose of 5mg/day. The option of considering a lower dose to the one currently considered as "standard" (10mg/day) is to reduce toxicity, mainly hematologic, in patients who do not receive treatment normally. A dose with lower toxicity has been chosen which has revealed itself efficient.

Main efficiency objective:

•To assess if treatment with Revlimid (Lenalidomide) extends the period until the progression to myelodysplastic syndrome del(5q) considered as transfusion independent, documented verification that the patient suffering from anemia due to MDS requires transfusion of at least 2 UCH/56 days (2 months) with a minimum follow up of 112 days (4 months). Revlimid will be compared to the current standard treatment for patients with low risk myelodysplastic syndrome associated with the loss of 5qwithout transfusion dependent anemia, which is the therapeutic abstention and monitoring until its progression.

Secondary efficiency objectives:

* Erythroid response according to the Criteria of the myelodysplastic syndrome International Work Team 2006).
* Duration of the red blood cells transfusion independency (defined as the number of days elapsed between the randomization and the first transfusion after this period free of transfusions).
* Change of hemoglobin concentration (Hb) in relation to baseline levels of patients who show erythroid response.
* Variation in platelets absolute count in relation to baseline levels.
* Variation in neutrophils absolute count in relation to baseline levels.
* Cytogenetic response according to the Criteria of the myelodysplastic syndrome International Work Team.
* Bone marrow response according to the Criteria of the myelodysplastic syndrome International Work Team.
* To assess the safety and tolerance of the Lenalidomide scheme, measured according to the incidence of clinical and laboratory toxicity.
* Global survival, Event Free Survival and Rate of Transformation to Acute Leukemia.
* Time from diagnose to transfusion independence.

Main safety objective:

Safety (type, frequency and severity [Criteria of normal terminology of adverse reactions of the National Cancer Institute (NCI CTCAE) version 3.0] of adverse reactions (AR)and list of the AR with Lenalidomide.

Four of the sites of this Clinical Trial are member of the European Reference Network on Rare Hematological Diseases (ERN-EuroBloodNet) which is partially co-funded by the European Union within the framework of the Third Health Programme. "ERN-2016 - Framework Partnership Agreement 2017-2021." FPA 739541".

ELIGIBILITY:
Inclusion Criteria:

1. - The patient must, in the investigator's opinion, be able to comply with all the clinical trial requirements.
2. - The patient must voluntarily sign the informed consent form before undergoing any test of the trial that is not part of the normal patient care, and patient must be aware that he/she can withdraw from the trial at any time, without it ever affecting their future healthcare.
3. - Age > 18 years.
4. - The patient must be diagnosed with low risk MDS (low and intermediate-1 IPSS) associated with 5q deletion, either as an isolated abnormality or accompanied by other additional cytogenetic abnormalities.
5. - MDS Del(5q) with transfusion-independent anaemia (Hb ≤ 12 g/dL), and documented confirmation that no packed red blood cells transfusion due to the patient's underlying condition (MDS) has been received.
6. - The patient must have an ECOG performance status of ≤ 2.
7. - The patient must be able to comply with the scheduled study visits.
8. - Female patient with childbearing potential must*:

   * Understands the teratogenic risk of the study drug.
   * Commits herself to use two forms of effective birth control continuously, and is able to use them correctly, for the 4 weeks prior to starting treatment with the study drug, as well as during treatment with the study drug (including periods of dose interruption), and for up to 4 weeks after finishing treatment with the study drug, even if amenorrhoeic. This always applies, except in women who commit to continued complete sexual abstinence, as confirmed on a monthly basis.
   * The patient must understand that even if she is amenorrhoeic she must follow all the advice on effective contraception.
   * The patient must understand the possible consequences of pregnancy and the need to attend a healthcare service urgently in case there is a risk of pregnancy.
   * Agree to undergo a pregnancy test with a minimum sensitivity of 25 mIU/mL, under medical supervision, on the day of the study visit or during the 3 days prior to this visit, after using effective birth control for at least 4 weeks. This requirement also applies to women with childbearing potential who practice complete and continued sexual abstinence. The test must confirm that the patient is not pregnant at the time the treatment is initiated.
   * Agree to undergo a pregnancy test, under medical supervision, weekly for he first 28 days of treatment, and subsequently every 4 weeks, including a pregnancy test 4 weeks after finishing the study treatment, except in case of confirmed tubal ligation. This pregnancy test will be performed on the day of the study visit or during the 3 days prior to it. This requirement also applies to women with childbearing potential who practice complete and continued sexual abstinence.
9. - All male patients must:

   * Commit himself to the use of condoms throughout all the treatment with the study drug, including all periods of dose interruption, and up to one week after finishing the treatment if their partner is a woman with childbearing potential and does not use birth control methods.
   * Commit himself to not donate semen during treatment with the study drug and up to one week after finishing the treatment.
10. - All patients must:

    * Refrain from donating blood while receiving treatment with the study drug and during the week following the end of the treatment.
    * Refrain from sharing the study drug with others, and return all unused study drug to the investigator or pharmacist.

Exclusion Criteria:

1. - Any organic disease or psychiatric disorder which makes it impossible for the patient to sign or understand the informed consent.
2. - Having received any treatment for MDS.
3. - Del(5q) MDS with transfusion-dependent anaemia, and documented confirmation that the patient has received any pRBC transfusion due to the underlying condition (MDS).
4. - Pregnant or breast-feeding women.
5. - Any of the following laboratory abnormalities:

   * Absolute neutrophil count < 500/mm3
   * Platelet count < 25,000/mm3
   * Serum GOT or GPT > 3 times the upper limit of normal values.
   * Total serum bilirubin > 2 times the upper limit of normal values.
6. - Previous history of other malignancies other than MDS (except for basal cell or squamous cell skin carcinoma, or carcinoma in situ of the cervix or breast), unless the patient has been free of disease for more than 5 years.
7. - Known hypersensitivity to or a history of uncontrollable side effects to lenalidomide.
8. - Major surgery within the 4 weeks prior to the inclusion in the trial.
9. - The patient has received any investigational agent in the 30 days prior to inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2010-01; Primary Completion 2022-06-06 (Actual); Study Completion 2022-06-06 (Actual)

PRIMARY OUTCOMES:
Period until the progression of myelodysplastic syndrome | 6 years (study treatment and follow up)
  To assess if treatment with Revlimid (Lenalidomide) extends the period until the progression to MDS of(5q) considered as transfusion independent, documented verification that the patient suffering from anemia due to MDS requires transfusion of at least 2 UCH/56 days (2 months) with a minimum follow up of 112 days (4 months). Revlimid will be compared to the current standard treatment for patients with low risk MDS associated with the loss of 5q without transfusion dependent anemia, which is the therapeutic abstention and monitoring until its progression.

SECONDARY OUTCOMES:
Erythroid response | 6 years (study treatment and follow up)
  Erythroid response according to the Criteria of the MDS International Work Team.
Duration of the red blood cells transfusion independency | 6 years (study treatment and follow up)
  Red blood cells transfusion independency,defined as the number of days elapsed between the randomization and the first transfusion after this period free of transfusions.
Change of the hemoglobin concentration (Hb) in relation to baseline levels | 6 years (study treatment and follow up)
  Change of the hemoglobin concentration (Hb) in relation to baseline levels of patients who show erythroid response.
Variation in platelets and neutrophils absolute count in relation to baseline levels | 6 years (study treatment and follow up)
  Variation in platelets and neutrophils absolute count in relation to baseline levels
Cytogenetic response | 6 years (study treatment and follow up)
  Cytogenetic response according to the Criteria of the MDS International Work Team.
Bone marrow response | 6 years (study treatment and follow up)
  Bone marrow response according to the Criteria of the MDS International Work Team.
Global survival, Event Free Survival and Rate of Transformation to Acute Leukemia. | 6 years (study treatment and follow up)
  Global survival, Event Free Survival and Rate of Transformation to Acute Leukemia
Time from diagnose to transfusion independence. | 6 years (study treatment and follow up)
  Time from diagnose to transfusion independence
Safety( type, frequency and severity of adverse events and relationship to lenalidomide | 6 years (study treatment and follow up)
  Safety (type, frequency and severity [Criteria of normal terminology of adverse reactions of the National Cancer Institute (NCI CTCAE) version 3.0] of adverse reactions (AR)and list of the AR with Lenalidomide.

CONTACTS AND LOCATIONS:
Overall Officials: Consuelo del Cañizo, MD, Study Chair — Hospital Clínico Universitario de Salamanca; María Díez Campelo, MD, Study Chair — Hospital Clínico Universitario de Salamanca
Locations (25):
- France (7):
  - Hôpitaux Universitaires de Strasbourg, Strasbourg, Bajo Rin
  - Centre Hospitalier Universitaire de Nîmes, Nîmes, Gard
  - Centre Hospitalier Régional d'Orléans, Orléans, Loiret
  - Centre Hospitalier Universitaire d'Angers, Angers, Maine Y Loira
  - Centre Hospitalier Universitaire Brabois, Nancy, Meurthe Y Mosel
  - Centre Hospitalier d'Avignon, Avignon, Vaucluse
  - Hôspital St. Louis, Paris
- Germany (3):
  - Universitaetsklinikum Carl Gustav Carus der Technischen Universitaet Dresden, Dresden
  - Marien Hospital Duesseldorf, Düsseldorf
  - Klinikum rechts der Isar der Technischen Universität München, München
- Spain (15):
  - Hospital Son Llàtzer, Palma de Mallorca, Balearic Islands
  - Hospital Universitari Germans Trias i Pujol (ICO Badalona), Badalona, Barcelona
  - Hospital de Cabueñes, Gijón, Principality of Asturias
  - Hospital Central de Asturias, Oviedo, Principality of Asturias
  - Hospital de Cruces, Barakaldo, Vizcaya
  - Hospital Clínic i Provincial, Barcelona
  - Hospital Universitario Reina Sofía, Córdoba
  - Instituto Catalán de Oncología de Gerona, Girona
  - Hospital Infanta Leonor, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital General Universitario José Maria Morales Meseguer, Murcia
  - Hospital Clínico Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario La Fe, Valencia

REFERENCES:
- [Background] Steensma DP, Tefferi A. The myelodysplastic syndrome(s): a perspective and review highlighting current controversies. Leuk Res. 2003 Feb;27(2):95-120. doi: 10.1016/s0145-2126(02)00098-x. PMID 12526916
- [Background] Greenberg P, Cox C, LeBeau MM, Fenaux P, Morel P, Sanz G, Sanz M, Vallespi T, Hamblin T, Oscier D, Ohyashiki K, Toyama K, Aul C, Mufti G, Bennett J. International scoring system for evaluating prognosis in myelodysplastic syndromes. Blood. 1997 Mar 15;89(6):2079-88. PMID 9058730
- [Background] List AF. New approaches to the treatment of myelodysplasia. Oncologist. 2002;7 Suppl 1:39-49. doi: 10.1634/theoncologist.7-suppl_1-39. PMID 11961208
- [Background] McHugh SM, Deighton J, Stewart AG, Lachmann PJ, Ewan PW. Bee venom immunotherapy induces a shift in cytokine responses from a TH-2 to a TH-1 dominant pattern: comparison of rush and conventional immunotherapy. Clin Exp Allergy. 1995 Sep;25(9):828-38. doi: 10.1111/j.1365-2222.1995.tb00025.x. PMID 8564721
- [Background] Bellamy WT. Expression of vascular endothelial growth factor and its receptors in multiple myeloma and other hematopoietic malignancies. Semin Oncol. 2001 Dec;28(6):551-9. doi: 10.1016/s0093-7754(01)90023-5. PMID 11740808
- [Background] Bartlett JB, Dredge K, Dalgleish AG. The evolution of thalidomide and its IMiD derivatives as anticancer agents. Nat Rev Cancer. 2004 Apr;4(4):314-22. doi: 10.1038/nrc1323. No abstract available. PMID 15057291
- [Background] List A, Kurtin S, Roe DJ, Buresh A, Mahadevan D, Fuchs D, Rimsza L, Heaton R, Knight R, Zeldis JB. Efficacy of lenalidomide in myelodysplastic syndromes. N Engl J Med. 2005 Feb 10;352(6):549-57. doi: 10.1056/NEJMoa041668. PMID 15703420
- [Background] List A, Dewald G, Bennett J, Giagounidis A, Raza A, Feldman E, Powell B, Greenberg P, Thomas D, Stone R, Reeder C, Wride K, Patin J, Schmidt M, Zeldis J, Knight R; Myelodysplastic Syndrome-003 Study Investigators. Lenalidomide in the myelodysplastic syndrome with chromosome 5q deletion. N Engl J Med. 2006 Oct 5;355(14):1456-65. doi: 10.1056/NEJMoa061292. PMID 17021321
- [Background] List A, Gordon W, Dewald G, Bennett J, Giagounidis A, Raza A et al. Long-term clinical benefit of lenalidomide (Revlimid) treatment in patients with myelodysplastic syndrome and chromosome deletion 5q [Abstract]. Blood. 2006;108:251A.
- [Background] Mallo M, Cervera J et al. Prognostic impact of additional chromosomal aberrations to 5q- in patients with primary myelodysplastic syndromes. Oral comunication, 0906, 13th Congress of the European Hematology Association. Haematologica | 2008; 93(s1), pag. 360
- [Background] Fenaux P, Kelaidi C. Treatment of the 5q- syndrome. Hematology Am Soc Hematol Educ Program. 2006:192-8. doi: 10.1182/asheducation-2006.1.192. PMID 17124060
- [Background] Kelaidi C, Eclache V, Fenaux P. The role of lenalidomide in the management of myelodysplasia with del 5q. Br J Haematol. 2008 Feb;140(3):267-78. doi: 10.1111/j.1365-2141.2007.06910.x. PMID 18217896
- [Background] List, AF. Active treatment-improving outcomes in del 5q patients. Leukemia Research, (2007)31(Suppl. 1), S9.
- [Derived] Diez-Campelo M, Lopez-Cadenas F, Xicoy B, Lumbreras E, Gonzalez T, Del Rey Gonzalez M, Sanchez-Garcia J, Coll Jorda R, Slama B, Hernandez-Rivas JA, Thepot S, Bernal T, Guerci-Bresler A, Bargay J, Amigo ML, Preudhomme C, Fenwarth L, Platzbecker U, Gotze KS, Arar A, Toribio S, Del Canizo C, Hernandez-Rivas JM, Fenaux P. Low dose lenalidomide versus placebo in non-transfusion dependent patients with low risk, del(5q) myelodysplastic syndromes (SintraREV): a randomised, double-blind, phase 3 trial. Lancet Haematol. 2024 Sep;11(9):e659-e670. doi: 10.1016/S2352-3026(24)00142-X. Epub 2024 Jul 18. PMID 39033767